CLINICAL TRIAL: NCT04981561
Title: A Phase 1, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AGN-241751 After Oral Administration in Healthy Volunteers
Brief Title: Safety and Tolerability of GATE-251 in Normal Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald M Burch MD PhD (Industry)
Responsible Party: Sponsor-Investigator, Ronald M Burch MD PhD, Chief Medical Officer, Syndeio Biosciences, Inc
Organization: Syndeio Biosciences, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3125-101-009
Record Dates: First submitted 2021-07-18; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
Keywords: NMDA receptor; NMDA receptor positive allosteric modulator; pharmacokinetics; biomarker; eeg
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 100 microgram GATE-251 (Experimental): GATE-251, 100 microgram tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 1 mg GATE-251 (Experimental): GATE-251, 1 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 3 mg GATE-251 (Experimental): GATE-251, 3 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 10 mg GATE-251 (Experimental): GATE-251, 10 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 25 mg GATE-251 (Experimental): GATE-251, 25 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 50 mg GATE-251 (Experimental): GATE-251, 50 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 100 mg GATE-251 (Experimental): GATE-251, 100 mg tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: GATE-251
- 1 mg GATE-251 with CSF collection (Experimental): GATE-251, 1 mg tablet, PO, Single Dose with 28 day follow up, with CSF collection
  Interventions: Drug: GATE-251
- 10 mg GATE-251 with CSF collection (Experimental): GATE-251, 10 mg tablet, PO, Single Dose with 28 day follow up, with CSF collection
  Interventions: Drug: GATE-251
- Placebo (Placebo Comparator): Placebo tablet, PO, Single Dose with 28 day follow up
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GATE-251 — Single dose of GATE-251
  Arms: 1 mg GATE-251; 1 mg GATE-251 with CSF collection; 10 mg GATE-251; 10 mg GATE-251 with CSF collection; 100 mg GATE-251; 100 microgram GATE-251; 25 mg GATE-251; 3 mg GATE-251; 50 mg GATE-251
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of single ascending doses of GATE-251 in normal human volunteers

DETAILED DESCRIPTION:
Single ascending dose (SAD), double-blind placebo-controlled study in normal human volunteers.

Secondary objectives:

To evaluate the pharmacokinetics (PK) and eeg biomarker of target engagement of GATE-251 following increasing single doses of GATE-251.

GATE-251 or Placebo: Dose/Mode of Administration: Single dose; oral

ELIGIBILITY:
Inclusion Criteria:

* Agree to effective method of birth control
* If female, negative pregnancy test at screening and Day -1
* Nonsmoking at least 2 years
* BMI 18-30
* Supine pulse rate 30-100

Exclusion Criteria:

* Known hypersensitivity to NMDA receptor drugs
* clinically significant disease in any body system
* QTcF > 430 ms in males, >450 ms in females
* positive test for hepatitis B or C
* abnormal liver function tests on Day -1
* History of alcohol or other substance abuse during the previous 5 years
* Positive drug screen at screening or Day -1
* Taken any medication within the past 14 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | 28 days
  through study completion

SECONDARY OUTCOMES:
Pharmacokinetics, maximum plasma concentration | 24 hours
  maximum plasma concentration
Pharmacokinetics, time to maximum plasma concentration | 24 hours
  time to maximum plasma concentration
Pharmacokinetics, area under the curve for plasma concentration | 72 hours
  area under the curve, plasma calculated 0-infinity

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD PhD, Study Director — Syndeio Biosciences, Inc